CLINICAL TRIAL: NCT07130552
Title: Comparison of Distal IPACK and Popliteal Plexus Block Combined With Femoral Triangle Block After Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-2022/16
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-06

CONDITIONS: Osteo Arthritis of the Knee
Keywords: Total knee arthroplasty; popliteal plexus block; femoral triangle block; iPACK block (infiltration of the interspace between the popliteal artery and the posterior knee capsule)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Popliteal plexus block (Experimental): femoral triangle block and popliteal plexus block
  Interventions: Device: femoral triangle block and popliteal plexus block
- Group distal iPACK (Experimental): Femoral triangle block and distal iPACK
  Interventions: Device: Femoral triangle block and distal iPACK

INTERVENTIONS:
Device: femoral triangle block and popliteal plexus block — Single dose bolus, 10 ml 5% bupivacaine will be used for FTB, 10 ml 5% bupivacaine will be used for PPB
  Arms: Group Popliteal plexus block
Device: Femoral triangle block and distal iPACK — Single dose bolus, 10 ml 5% bupivacaine will be used for FTB, 10 ml 5% bupivacaine will be used for distal iPACK
  Arms: Group distal iPACK

SUMMARY:
This study aims to investigate the effect of femoral triangle block combined with popliteal plexus block and distal IPACK block on postoperative pain after total knee arthroplasty (TKA)

DETAILED DESCRIPTION:
Popliteal Plexus Block (PPB) is a new nerve block technique that has been shown to anaesthetise nerves involved in the innervation of the posterior part of the knee joint.

The IPACK (interspace between the popliteal artery and capsule of the posterior knee) block is a regional anesthesia technique in which a local anesthetic is infiltrated under ultrasound guidance between the popliteal artery and the capsule of the posterior knee. This technique blocks the branches of the obturator nerve, the common peroneal nerve, and the tibial nerve in the popliteal region. In the context of knee arthroplasty, the application of the IPACK block has been associated with lower scores for ambulatory pain, lower scores for resting pain, and reduced morphine consumption.

Although both techniques of blockade seem to be efficient in the context of analgesia for the posterior part of the knee after TKA. No study compares these two blocks as part of multimodal analgesia to provide pain relief after TKA.

This study aimed to evaluate the analgesic effect of PPB or distal IPACK, in addition to femoral triangle block, as a component of a multimodal analgesic regimen after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee arthroplasty under spinal anesthesia
* American Society of Anesthesiologists (ASA) status I-III
* Patients who give informed consent

Exclusion Criteria:

* Patients unable to cooperate
* Kidney disease with GFR < 50 ml/min
* Daily opioid consumption > 1 month
* Allergy to local anesthetics
* Neurological problems of the lower extremity
* Contraindications to peripheral nerve blocks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 Years and older (Adult, Older Adult)
Enrollment: 120 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours
  Total opioid consumption in each group, A, B until 24 hours postoperative.

SECONDARY OUTCOMES:
NRS scores | 48 hours
  Numerical Rating Scale (NRS) scores (Range 0-10, 0=no pain, 10=the worse pain ever)
Range of knee motion | 48 hours
  Degrees of flexion
Patient mobilization | 48 hours
  Patient reporting time of first standing to the side of the bed and time up and go test 2 days
Post-block Maximum Voluntary Isometric Contraction (MVIC) by knee extension, calculated as a percentage of the Pre-block baseline value | A 60-minute interval is between pre-block and post-block MVIC assessments
  Both MVIC test are assessed preoperative, using a handheld dynamometer
Post-block MVIC by ankle plantarflexion, calculated as a percentage of the Pre-block baseline value | A 60-minute interval is between pre-block and post-block MVIC assessments
  Both MVIC tests are assessed preoperative, using a handheld dynamometer
Post-block MVIC by ankle dorsiflexion, calculated as a percentage of the Pre-block baseline value | A 60 minutes interval is between pre-block and post-block MVIC assessments
  Both MVIC tests are assessed preoperative, using a handheld dynamometer
Muscle strength of knee extension, graded by Manual Muscle Test (MMT) | Assessed pre-block, post-block (60 minutes after pre-block), and postoperative 5 hours
  Grade 3: Able to extend the knee in active Range of Motion (ROM) against gravity, Grade 2: Patient is lying on the side, with knee resting on the bed, able to extend the knee in active ROM with minimal assistance from the investigator, Grade 1: Muscle contraction of the quadriceps muscle is palpable or observable but the knee does not extend, Grade 0: No muscle contraction of the quadriceps muscle is palpable or observable
Muscle strength of ankle plantarflexion, graded by MMT | Assessed pre-block, post-block (60 minutes after pre-block) and postoperative 5 hours
  Grade 3: Able to plantarflex in active ROM, Grade 2: Patient is lying on the side, with ankle resting on the bed, able to plantarflex the ankle in active ROM with minimal assistance from the investigator, Grade 1: Muscle contraction of the gastrocnemius muscle is palpable or observable but the ankle does not plantarflex, Grade 0: No muscle contraction of the gastrocnemius muscle is palpable or observable
Muscle strength of ankle dorsiflexion, graded by MMT | Assessed pre-block, post-block (60 minutes after pre-block) and postoperative 5 hours
  Grade 3: Able to dorsiflex in active ROM Grade 2: Patient is lying on the side, with ankle resting on the bed, able to dorsiflex the ankle in active ROM with minimal assistance from the investigator, Grade 1: Muscle contraction of the tibialis anterior muscle is palpable or observable but the ankle does not dorsiflex, Grade 0: No muscle contraction of the tibialis anterior muscle is palpable or observable
Incidence of rebound pain | Postoperative 24 hours
  Rebound pain is described as severe pain (NRS ≥ 7)
Quality of Recovery 15 Score | Postoperative Day 1
  Quality of Recovery (QoR)-15 survey.Minimum value: 0, Maximum value: 150, higher scores mean better.

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman Training and Research Hospital, Karaman, Karaman 70200, Karaman, Karaman, Turkey (Türkiye)